CLINICAL TRIAL: NCT04779567
Title: Randomized Double-blind Controlled Study to Assess the Efficacy of Intravenous Acetaminophen Associated With Strong Opioids in the Management of Acute Pain in Adult Cancer Patients
Brief Title: Usefulness of Acetaminophen Associated With Strong Opioids for Acute Pain in Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 180328004
Record Dates: First submitted 2020-11-18; First posted 2021-03-03 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-06

CONDITIONS: Acute Pain; Cancer Pain
MeSH Terms: conditions — Acute Pain; Cancer Pain | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: Prospective, Single center parallel-group, randomized double-blinded controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: matching placebo. prepared by pharmacist
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen (Experimental): Acetaminophen 1 gr in 100 ml saline 0,9% iv 4 times a day
  Interventions: Drug: Acetaminophen
- Placebo (Placebo Comparator): 100 ml saline 0.9% iv 4 times a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen 1 gr iv 4 times a day
  Arms: Acetaminophen
Drug: Placebo — 100 ml saline 0.9% iv 4 times a day
  Arms: Placebo

SUMMARY:
Cancer pain is one of the most frequent and relevant symptoms in cancer patients and has a great impact on a patient's quality of life. International and local standards recommend as an initial strategy, the use of an analgesic scheme composed of strong opioids (morphine, methadone or fentanyl) associated with adjuvants such as paracetamol, based upon the assumption that the use of combined analgesics could have a better analgesic effect, could allow the use of lower dose of opioids and that also could prevent the occurrence of adverse effects of opioids. However, there is uncertainty about the impact of paracetamol as an adjuvant in patients who use strong opioids for pain management in cancer patients with moderate to severe pain.

To clarify this question, this study aims to evaluate the efficacy and safety of intravenous paracetamol associated with strong opioids in hospitalized cancer patients who have pain associated with cancer of moderate to severe intensity, (4 or more), older than 18 years.

Randomized double-blinded controlled study comparing intravenous acetaminophen 1 gr 4 times a day versus placebo for 48 hours as an adjuvant to strong opioids. We will assess pain intensity as a primary outcome validated assessments that estimate Verbal Numerical Rating Scale (VNRS) analogous verbal pain from 0 to 10, and de visual Analog Scale (VAS). We estimated that a decrease of 1 point on the verbal numerical scale would be statistically significant. In addition, the investigators will calculate the amount of total opioid dose in 24 hours and then perform the intervention. As a secondary outcome, adverse effects such as drowsiness, constipation, nausea and vomiting would be evaluated

DETAILED DESCRIPTION:
This is a randomized, controlled, double blind, parallel-group, single center clinical trial. This study received ethical approval by the Ethics Committee of the Pontificia Universidad Católica de Chile (ID #180328004). The study protocol was designed using the recommendations of the Consolidated Standards of Reporting Trials (CONSORT) statement.

The setting of this study is the General Internal Medicine Ward of a tertiary level university hospital (UC Christus Clinical Hospital) where patients will be recruited.

The hypothesis of this study is that in hospitalized oncology patients over 18 years of age, acute pain management with strong opioids plus intravenous paracetamol is not superior to the use of strong opioids alone.

Participants Patients 18 years old or older, diagnosed with cancer and admitted to UC Christus Clinical Hospital of any ethnicity or nationality with moderate to severe pain.All participate in the study will sign an informed consent form.

Treatments Opioid administration - Before starting the study a standardized pain management protocol for cancer patients with moderate to severe pain will be implemented across the institution. In this protocol, a standard analgesic protocol (scheduled strong opioids plus rescue doses, such as morphine, methadone or fentanyl) will be started by the ward team upon admission in order to ensure that all cancer patients with moderate to severe pain will have an adequate analgesic scheme for pain control regardless study enrollment. Briefly, cancer patients with moderate to severe pain who are opioid naive will be started on scheduled morphine, methadone or fentanyl by continuous infusion plus rescue doses. Standard doses will be recommended but these doses could be changed by treating clinicians according to clinical judgement. For patients with prior use of opioids, ward or treating clinicians could start scheduled methadone or morphine or fentanyl continuous infusion increasing the prior opioid dose. Early consultation to palliative care clinicians will be recommended for this population.

Acetaminophen - experimental group - Intravenous acetaminophen is usually delivered in a 100cc solution that is prepared in a transparent glass bottle. As the placebo cannot be prepared in the same type of bottle, the content of the acetaminophen preparation will be transferred to a standard 100cc plastic flask for IV infusions, which will be labeled with the name and ID number of the patient, with the drug to be administered labeled acetaminophen/placebo (including both names) and with the allocation number for the randomization. The preparation of the acetaminophen plastic flask will be indistinguishable from the placebo plastic flask. As the intervention will last 48 hours, 8 plastic flasks with the drug will be sent directly to the clinical nurse in charge of the administration of the drug in the general ward.

Placebo - control group - The placebo will be prepared using the same plastic flask as used in the acetaminophen group. In the placebo group it will be filled with 100cc of saline, and will have the same label as the acetaminophen group, therefore they will be indistinguishable from each other. In the case of the placebo group, 8 plastic flasks with the placebo will be sent directly to the clinical nurse in charge of the administration of the drug in the general ward.

Other treatments - As the research group wants to assess the impact of this intervention in the real clinical setting, treating clinicians will be allowed to be added according to clinical judgement. Non-steroidal anti inflammatories (NSAIDS), steroids, anticonvulsants, or other adjuvants could be added.

Randomization - After informed consent, eligible patients will be randomized into two arms: (A) acetaminophen or (B) placebo. The randomization procedure will be performed by the institution's pharmacist using a web-based randomization software platform specifically designed to support data collection for research studies (Research Electronic Data Capture, REDCap®), platform that provides automated export procedures for data downloads. The randomization will be performed following a stratified block randomization, with blocks of 4 or 6 patients among which 50% of each block will receive placebo and 50% will receive acetaminophen. The study will be blind with randomization concealment. Once the pharmacist has identified the allocated arm of the enrolled patient, a total of 8 identical plastic flasks will be prepared in the pharmacy service, with a total amount of 100ml of volume each and each one labeled as previously described. For arm (A), IV acetaminophen will be prepared, for arm (B), IV saline will be prepared. The eight plastic flasks will be delivered to the general ward and the clinical nurses will be in charge of administering the infusions during the 48 hours study period. Precautions will be taken to ensure that treating physicians, clinical nurses, data collectors, data adjudicators, patients and researchers will be blind to patient allocation.

Follow-up and data collection - Patients will be asked to complete a baseline assessment questionnaire and then two other questionnaires at 24 and 48 hours after enrollment. The questionnaires were selected seeking to assess the primary and secondary outcomes and variables that could impact patients' pain experience. We included a variety of questionnaires and instruments, to assess eligibility criteria, the primary and secondary outcomes and possible affect modifiers, including instruments to assess delirium (Memorial Delirium [MDAS]), pain (Verbal Numerical Rating Scale [VNRS] and Visual Analog Scale [VAS]), use of analgesia prior to admission, alcohol and drug consumption, risk of chemical coping, symptoms, psychological distress (Hospital Anxiety Depression Scale [HADS]), quality of life and symptoms associated with their current hospitalization .

Data collection and management Sample size - To estimate the sample size, we decided to use the strategy of identifying the minimum clinically important difference (MCID) in pain according to the ESAS scale, which evaluates pain on a scale from 0 to 10, similar to the VNRS, which we will use as our main outcome. The MCID is defined as "the smallest change in a measurement that signifies an important difference in a patient's symptoms". In a study conducted by Farrar, et al, the MCID for pain was defined as 2 points, which was evaluated in a short in-hospital follow-up period, a scenario that is similar to that of our study. In another study, conducted by Hui, et al , published in 2015, different methods for establishing MCID were evaluated. In that study, using the anchor-based method through the calculation of the ROC curve, it was recognized that an improvement in pain intensity by 1 point on the ESAS scale was identified by patients as a clinically significant improvement, i.e. patients detect 1 point on the ESAS scale as an improvement in pain control, scale similar to the VNRS. In this study the standard deviation for the pain score was 3 points, similarly to what was found in previous studies. Using other similar strategies, a difference between 1 and 2 points was identified as clinically significant. However, in this study the pain assessment was performed on an outpatient basis and with a 3-week difference between the first and the last assessment.

In an unpublished sample of 100 advanced cancer patients assessed in our PC unit, we found that the mean intensity of pain using the VNRS among patients with moderate to severe pain was 5,8 points with a standard deviation (SD) of 1.7 points.

From the data obtained from prior publications, considering an alpha of 0.025, with a power of 0.8, we estimated that a sample size 112 patients would be required, with 56 patients in each group to detect a difference of 1 point in pain intensity between the groups, with a standard deviation (SD) of 1.7. These assumptions are supported by the following reasons:

Because a difference of 1 point is considered to be what is clinically defined as significant, so we should try to detect a difference greater than that.

Because we reported an SD of 1.7 in the initial pain scale in a sample of cancer patients in our unit.

In this way the investigators could be able to recommend, not to use intravenous paracetamol, which would generate an indirect recommendation not to use oral paracetamol in patients with moderate to severe acute pain associated with cancer. This not only has an economic impact, but also could affect the well-being of patients who are sometimes in a great pharmacological burden, in the context of low oral intake and frequent nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients hospitalized at UC Christus Clinical Hospital of any ethnicity or nationality.
* With acute pain> or = a 4 in Verbal Numerical Rating Scale (VNRS)
* They can be patients who are virgins to opioids or previous users of weak or strong opioids.
* They may have somatic, visceral or neuropathic pain
* They may be users of NSAIDs or corticosteroids

Exclusion Criteria:

* Patients who refuse to enter the study
* Patients who don´t speak Spanish a mother language
* Patients who present a qualitative or quantitative awareness commitment that prevents the assessment of pain.
* Patients with acute liver failure or chronic liver damage Child C.
* Patients allergic or hypersensitive to paracetamol.
* Patients with a prognosis of life less than 72 hours (evaluated according to clinical criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Efficacy of acetaminophen by Verbal Numerical Rating Scale (VNRS) | 48 hours
  The primary outcome of this study will be the difference in pain intensity between baseline (T=0) and 48 hours (T=2) using the Verbal Numerical Rating Scale (VNRS) reported by the patient to assess the effects of the intervention in pain intensity. We will compare the difference in pain intensity between the groups. The VNRS is a tool in which the patient is asked to score the mean intensity of pain during the last 24 hours in a scale from 0 to 10 with 0 meaning no pain at all and 10 meaning the worst possible pain.
Efficacy of acetaminophen by Visual Analog scale (VAS), in a scale from 0 to 10 with 0 meaning no pain at all and 10 meaning the worst possible pain. | 48 hours
  The VAS uses a right triangle drawn on a paper, with a base of 10 cm wide and a height of 1cm on the right, in which its ends are delimited by a mark that expresses "without pain" on the left side and" worst pain I have ever felt" on the right side. The patient is asked to mark a vertical line crossing the horizontal line indicating the intensity of the pain. On the reverse, there is a superimposed line, with a graduation of 1 cm wide, which allows the data collector to identify the position in which the line marked by the patient is located. This indicates patients´ pain intensity score assigned by the patient on a scale from 0 to 10. We will also estimate the difference in pain intensity between baseline and 48 hours using the VAS and compare the magnitude of the difference between the arms.
Efficacy of acetaminophen by total morphine equivalent daily dose (MEDD) | 48 Hours
  MEDD at 48 hours. The MEDD represents the total dose of opioids used within the last 24 hours converted into an equivalent dose of parenteral morphine, following standard equianalgesic conversion tables

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | T1: 24 hours and T2: 48 Hours
  Incidence of treatment-emergent adverse Events: Drowsiness, constipation, nausea and vomit, allergy reactions.The patient is asked if he has presented any adverse effect to the treatment and this is classified as mild, moderate and severe

CONTACTS AND LOCATIONS:
Overall Officials: Ofelia Leiva, MD, Study Director — Universidad Católica de Chile
Locations (1):
- Universidad Catolica de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Yes
For numerical variables, baseline characteristic data were analyzed and represented with mean±SD, or median with interquartile range (IQR), according to data type and distribution. Categorical variables are presented as frequency and percentage.
  For bivariate analysis, Student T-test or ANOVA were used for enough sample size to assume Normal distribution of the averages by Central Limit Theorem, and Wilcoxon's rank sum test for non-normal distribution data.
  Finally, multivariate mixed models will be adjusted for interest scores: VAS, VNRS and MEEDs at 48 hours. As fixed effects in the model, we will consider de intervention (placebo or paracetamol) and other factors (as tabacco) and the patient as the random effect. A significance of 0.05 will be considered. The analyzes will be performed using the statistical package STATA 14.0.
Supporting Information: Study Protocol
Time Frame: We are unable to make the data available in a public repository or uploaded as supplementary information because this is not permitted by our organisation's research governance policy and Ethics committee regulations. Anonymised data can be made available to researchers who meet the conditions of the ethics approval and research governance policy that applies to this study. Researchers may request anonymized data access by contacting Universidad Católica's School of Medicine Research Office (DIDEMUC) at didemuc@med.puc.cl.

REFERENCES:
- [Result] van den Beuken-van Everdingen MHJ, de Rijke JM, Kessels AG, Schouten HC, van Kleef M, Patijn J. High prevalence of pain in patients with cancer in a large population-based study in The Netherlands. Pain. 2007 Dec 5;132(3):312-320. doi: 10.1016/j.pain.2007.08.022. Epub 2007 Oct 3. PMID 17916403
- [Result] Teunissen SC, Wesker W, Kruitwagen C, de Haes HC, Voest EE, de Graeff A. Symptom prevalence in patients with incurable cancer: a systematic review. J Pain Symptom Manage. 2007 Jul;34(1):94-104. doi: 10.1016/j.jpainsymman.2006.10.015. Epub 2007 May 23. PMID 17509812
- [Result] Goudas LC, Bloch R, Gialeli-Goudas M, Lau J, Carr DB. The epidemiology of cancer pain. Cancer Invest. 2005;23(2):182-90. PMID 15813511
- [Result] Portenoy RK, Ahmed E. Principles of opioid use in cancer pain. J Clin Oncol. 2014 Jun 1;32(16):1662-70. doi: 10.1200/JCO.2013.52.5188. Epub 2014 May 5. PMID 24799466
- [Result] Jimenez de la Jara J, Bastias G, Ferreccio C, Moscoso C, Sagues S, Cid C, Bronstein E, Herrera C, Nervi B, Corvalan A, Velasquez EV, Gonzalez P, Castellon E, Bustamante E, Onate S, McNerney E, Sullivan R, Owen GI. A snapshot of cancer in Chile: analytical frameworks for developing a cancer policy. Biol Res. 2015 Jan 26;48(1):10. doi: 10.1186/0717-6287-48-10. PMID 25761441
- [Result] Hui D, Bruera E. A personalized approach to assessing and managing pain in patients with cancer. J Clin Oncol. 2014 Jun 1;32(16):1640-6. doi: 10.1200/JCO.2013.52.2508. Epub 2014 May 5. PMID 24799495
- [Result] Johnston M, Pollard B, Hennessey P. Construct validation of the hospital anxiety and depression scale with clinical populations. J Psychosom Res. 2000 Jun;48(6):579-84. doi: 10.1016/s0022-3999(00)00102-1. PMID 11033377
- [Result] Chang VT, Hwang SS, Feuerman M. Validation of the Edmonton Symptom Assessment Scale. Cancer. 2000 May 1;88(9):2164-71. doi: 10.1002/(sici)1097-0142(20000501)88:93.0.co;2-5. PMID 10813730
- [Result] Delgado-Guay MO, Parsons HA, Hui D, De la Cruz MG, Thorney S, Bruera E. Spirituality, religiosity, and spiritual pain among caregivers of patients with advanced cancer. Am J Hosp Palliat Care. 2013 Aug;30(5):455-61. doi: 10.1177/1049909112458030. Epub 2012 Sep 4. PMID 22952129
- [Result] Latorres M, Huidobro A. [Prevalence of alcohol consumption among medical students at the Universidad Catolica del Maule, Chile]. Rev Med Chil. 2012 Sep;140(9):1140-4. doi: 10.4067/S0034-98872012000900006. Spanish. PMID 23354635
- [Result] Cleeland CS, Mendoza TR, Wang XS, Chou C, Harle MT, Morrissey M, Engstrom MC. Assessing symptom distress in cancer patients: the M.D. Anderson Symptom Inventory. Cancer. 2000 Oct 1;89(7):1634-46. doi: 10.1002/1097-0142(20001001)89:73.0.co;2-v. PMID 11013380
- [Result] Jadad AR, Browman GP. The WHO analgesic ladder for cancer pain management. Stepping up the quality of its evaluation. JAMA. 1995 Dec 20;274(23):1870-3. PMID 7500538
- [Result] Cherny N, Ripamonti C, Pereira J, Davis C, Fallon M, McQuay H, Mercadante S, Pasternak G, Ventafridda V; Expert Working Group of the European Association of Palliative Care Network. Strategies to manage the adverse effects of oral morphine: an evidence-based report. J Clin Oncol. 2001 May 1;19(9):2542-54. doi: 10.1200/JCO.2001.19.9.2542. PMID 11331334
- [Result] Barnes J, Abban M, Howarth P. Deaths from low dose paracetamol poisoning. Executive action is needed to change national guidelines. BMJ. 1998 Dec 12;317(7173):1654. No abstract available. PMID 9848918
- [Result] Toms L, McQuay HJ, Derry S, Moore RA. Single dose oral paracetamol (acetaminophen) for postoperative pain in adults. Cochrane Database Syst Rev. 2008 Oct 8;2008(4):CD004602. doi: 10.1002/14651858.CD004602.pub2. PMID 18843665
- [Result] McQuay HJ, Moore RA. Dose-response in direct comparisons of different doses of aspirin, ibuprofen and paracetamol (acetaminophen) in analgesic studies. Br J Clin Pharmacol. 2007 Mar;63(3):271-8. doi: 10.1111/j.1365-2125.2006.02723.x. Epub 2006 Jul 21. PMID 16869819
- [Result] Moore RA, Derry S, Wiffen PJ, Straube S, Aldington DJ. Overview review: Comparative efficacy of oral ibuprofen and paracetamol (acetaminophen) across acute and chronic pain conditions. Eur J Pain. 2015 Oct;19(9):1213-23. doi: 10.1002/ejp.649. Epub 2014 Dec 22. PMID 25530283
- [Result] Politi JR, Davis RL 2nd, Matrka AK. Randomized Prospective Trial Comparing the Use of Intravenous versus Oral Acetaminophen in Total Joint Arthroplasty. J Arthroplasty. 2017 Apr;32(4):1125-1127. doi: 10.1016/j.arth.2016.10.018. Epub 2016 Oct 21. PMID 27839957
- [Result] Hansen RN, Pham AT, Boing EA, Lovelace B, Wan GJ, Miller TE. Comparative analysis of length of stay, hospitalization costs, opioid use, and discharge status among spine surgery patients with postoperative pain management including intravenous versus oral acetaminophen. Curr Med Res Opin. 2017 May;33(5):943-948. doi: 10.1080/03007995.2017.1297702. Epub 2017 Mar 9. PMID 28276273
- [Result] Caraceni A, Hanks G, Kaasa S, Bennett MI, Brunelli C, Cherny N, Dale O, De Conno F, Fallon M, Hanna M, Haugen DF, Juhl G, King S, Klepstad P, Laugsand EA, Maltoni M, Mercadante S, Nabal M, Pigni A, Radbruch L, Reid C, Sjogren P, Stone PC, Tassinari D, Zeppetella G; European Palliative Care Research Collaborative (EPCRC); European Association for Palliative Care (EAPC). Use of opioid analgesics in the treatment of cancer pain: evidence-based recommendations from the EAPC. Lancet Oncol. 2012 Feb;13(2):e58-68. doi: 10.1016/S1470-2045(12)70040-2. PMID 22300860
- [Result] Vardy J, Agar M. Nonopioid drugs in the treatment of cancer pain. J Clin Oncol. 2014 Jun 1;32(16):1677-90. doi: 10.1200/JCO.2013.52.8356. Epub 2014 May 5. PMID 24799483
- [Result] Stockler M, Vardy J, Pillai A, Warr D. Acetaminophen (paracetamol) improves pain and well-being in people with advanced cancer already receiving a strong opioid regimen: a randomized, double-blind, placebo-controlled cross-over trial. J Clin Oncol. 2004 Aug 15;22(16):3389-94. doi: 10.1200/JCO.2004.09.122. PMID 15310785
- [Result] Axelsson B, Borup S. Is there an additive analgesic effect of paracetamol at step 3? A double-blind randomized controlled study. Palliat Med. 2003 Dec;17(8):724-5. doi: 10.1177/026921630301700816. No abstract available. PMID 14694929
- [Result] Israel FJ, Parker G, Charles M, Reymond L. Lack of benefit from paracetamol (acetaminophen) for palliative cancer patients requiring high-dose strong opioids: a randomized, double-blind, placebo-controlled, crossover trial. J Pain Symptom Manage. 2010 Mar;39(3):548-54. doi: 10.1016/j.jpainsymman.2009.07.008. Epub 2010 Jan 18. PMID 20083373
- [Result] Cubero DI, del Giglio A. Early switching from morphine to methadone is not improved by acetaminophen in the analgesia of oncologic patients: a prospective, randomized, double-blind, placebo-controlled study. Support Care Cancer. 2010 Feb;18(2):235-42. doi: 10.1007/s00520-009-0649-8. Epub 2009 May 7. PMID 19421788
- [Result] Tasmacioglu B, Aydinli I, Keskinbora K, Pekel AF, Salihoglu T, Sonsuz A. Effect of intravenous administration of paracetamol on morphine consumption in cancer pain control. Support Care Cancer. 2009 Dec;17(12):1475-81. doi: 10.1007/s00520-009-0612-8. Epub 2009 Apr 3. PMID 19343373
- [Result] Nabal M, Librada S, Redondo MJ, Pigni A, Brunelli C, Caraceni A. The role of paracetamol and nonsteroidal anti-inflammatory drugs in addition to WHO Step III opioids in the control of pain in advanced cancer. A systematic review of the literature. Palliat Med. 2012 Jun;26(4):305-12. doi: 10.1177/0269216311428528. Epub 2011 Nov 29. PMID 22126843
- [Result] Perez-Cruz PE, Padilla Perez O, Bonati P, Thomsen Parisi O, Tupper Satt L, Gonzalez Otaiza M, Ceballos Yanez D, Maldonado Morgado A. Validation of the Spanish Version of the Quality of Dying and Death Questionnaire (QODD-ESP) in a Home-Based Cancer Palliative Care Program and Development of the QODD-ESP-12. J Pain Symptom Manage. 2017 Jun;53(6):1042-1049.e3. doi: 10.1016/j.jpainsymman.2017.02.005. Epub 2017 Mar 16. PMID 28323080
- [Result] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Result] Hui D, dos Santos R, Chisholm G, Bansal S, Silva TB, Kilgore K, Crovador CS, Yu X, Swartz MD, Perez-Cruz PE, Leite Rde A, Nascimento MS, Reddy S, Seriaco F, Yennu S, Paiva CE, Dev R, Hall S, Fajardo J, Bruera E. Clinical signs of impending death in cancer patients. Oncologist. 2014 Jun;19(6):681-7. doi: 10.1634/theoncologist.2013-0457. Epub 2014 Apr 23. PMID 24760709
- [Result] Hui D, Shamieh O, Paiva CE, Perez-Cruz PE, Kwon JH, Muckaden MA, Park M, Yennu S, Kang JH, Bruera E. Minimal clinically important differences in the Edmonton Symptom Assessment Scale in cancer patients: A prospective, multicenter study. Cancer. 2015 Sep 1;121(17):3027-35. doi: 10.1002/cncr.29437. Epub 2015 Jun 8. PMID 26059846
- [Result] Farrar JT, Portenoy RK, Berlin JA, Kinman JL, Strom BL. Defining the clinically important difference in pain outcome measures. Pain. 2000 Dec 1;88(3):287-294. doi: 10.1016/S0304-3959(00)00339-0. PMID 11068116
- [Result] WHO Guidelines for the Pharmacological and Radiotherapeutic Management of Cancer Pain in Adults and Adolescents. Geneva: World Health Organization; 2018. Available from http://www.ncbi.nlm.nih.gov/books/NBK537492/ PMID 30776210
- [Result] Wiffen PJ, Derry S, Moore RA, McNicol ED, Bell RF, Carr DB, McIntyre M, Wee B. Oral paracetamol (acetaminophen) for cancer pain. Cochrane Database Syst Rev. 2017 Jul 12;7(7):CD012637. doi: 10.1002/14651858.CD012637.pub2. PMID 28700092
- [Derived] Leiva-Vasquez O, Letelier LM, Rojas L, Viviani P, Castellano J, Gonzalez A, Perez-Cruz PE. Is Acetaminophen Beneficial in Patients With Cancer Pain Who are on Strong Opioids? A Randomized Controlled Trial. J Pain Symptom Manage. 2023 Sep;66(3):183-192.e1. doi: 10.1016/j.jpainsymman.2023.05.002. Epub 2023 May 18. PMID 37207788
- [Derived] Leiva O, Castellano J, Letelier LM, Rojas L, Viviani P, Gonzalez A, Perez-Cruz P. Randomized double-blind controlled trial to assess the efficacy of intravenous acetaminophen associated with strong opioids in the treatment of acute pain in adult cancer patients: study protocol. Trials. 2022 Jul 6;23(1):548. doi: 10.1186/s13063-022-06442-2. PMID 35794673
- See also: Health Ministry — https://www.minsal.cl/portal/url/item/72213ed52c2723d1e04001011f011398.pdf
- See also: Cancer pain relief. With a Guide to opioid availability — https://apps.who.int/iris/bitstream/handle/10665/37896/9241544821.pdf;jsessionid=46F526101B59DBB6773822B1A44B3A5E?sequence=1
- See also: Palliative care guideline — http://www.who.int/cancer/palliative/painladder/en/

DOCUMENTS (1):
  • Informed Consent Form (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT04779567/ICF_000.pdf